CLINICAL TRIAL: NCT05197296
Title: Zooming in on Cerebral Abnormalities in Severely Affected COVID-19 Patients: a 3T and 7T MRI Study
Brief Title: Zooming in on Cerebral Abnormalities in Severely Affected COVID-19 Patients
Acronym: ZoomCOVID
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 79868
Record Dates: First submitted 2022-01-17; First posted 2022-01-19 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: COVID-19; Intensive Care Unit
Keywords: Magnetic Resonance Imaging; Intensive Care Unit; COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood (approximately 20mL in total) will be drawn using heparin, EDTA, serum and citrate tubes to evaluate markers for hypercoagulation and inflammation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brain injury is one of the complications in COVID-19 intensive care unit (ICU) survivors, though the precise underlying mechanism is unclear. It is likely caused by a combination of prolonged hypoxia, a massive systemic inflammatory response, direct infection of the brain and small vessel vasculitis in combination with widespread hypercoagulopathy and thrombosis. Using novel MRI techniques, blood-brain barrier (BBB) permeability, as well as other microstructural and microvascular properties of the brain tissue, will be assessed non-invasively in COVID-19 ICU survivors approximately one year after ICU admission and compared to serial clinical and laboratory measurements of hypercoagulation and inflammation during the (ICU) admission. This study aims to relate factors of hypercoagulability, inflammation or general illness itself (all during ICU admission) to microstructural and microvascular abnormalities on follow-up brain advanced 3T and 7T MRI in COVID-19 ICU survivors. In addition, neuropsychological tests and an objective smell/taste test will be used to evaluate neuropsychological status and sense of smell/taste. By gaining more insight into the pathogenesis of brain injury, the treatment of COVID-19 patients in the acute phase might be improved.

DETAILED DESCRIPTION:
Brain injury is one of the complications in COVID-19 intensive care unit (ICU) survivors, though the precise underlying mechanism is unclear. It is likely caused by a combination of prolonged hypoxia, a massive systemic inflammatory response, direct infection of the brain and small vessel vasculitis in combination with widespread hypercoagulopathy and thrombosis. Using novel MRI techniques, blood-brain barrier (BBB) permeability, as well as other microstructural and microvascular properties of the brain tissue, will be assessed non-invasively in COVID-19 ICU survivors approximately 12-24 months after ICU admission and compared to serial clinical and laboratory measurements of hypercoagulation and inflammation during the (ICU) admission.

This study aims to relate factors of hypercoagulability, inflammation or general illness itself (all during ICU admission) to microstructural and microvascular abnormalities on follow-up brain advanced 3T and 7T MRI in COVID-19 ICU survivors. By gaining more insight into the pathogenesis of brain injury, the treatment of COVID-19 patients in the acute phase might be improved.

This is a mono-center follow-up cohort study with measurements at 12-24 months post hospital discharge. This study will include 70 adults who survived a severe COVID-19 infection for whom ICU admission was necessary during the second/third COVID wave (period October 2020- ongoing). These patients will be recruited from the MaastrICCht cohort from the Department of Intensive Care (MUMC+).

Patients will undergo an MRI scan (3T) and optionally a second MRI scan (7T) of approximately 60 minutes each. These scans will lead to insights in microstructural and microvascular abnormalities, BBB impairment, and in possible effects of a severe COVID-19 infection on the brainstem and the glymphatic system. In addition to the MRI measurements, blood samples will be drawn (approximately 20ml) to evaluate ICU follow-up levels of hypercoagulation and inflammation biomarkers. Follow-up short neuropsychological tests and two short questionnaires will be used to assess cognitive, neurological, olfaction and functional status. A brief objective smell and taste testing will be done to get an objective measure of sense of smell and taste.

By gaining more insight into the pathogenesis of brain injury, the treatment of COVID-19 patients in the acute phase might be improved.

ELIGIBILITY:
Inclusion Criteria:

* Proven COVID-19 infection for which participant was admitted to the ICU for at least 3 days
* Included in the MaastrICCht cohort (a large database of serial measurements collected during ICU stay from patients with COVID-19 admitted to the ICU in the Maastricht University Medical Center+)
* Informed consent is given
* Sufficient command of the Dutch language to follow test instructions and understand the information letter, informed consent, and questionnaires

Exclusion Criteria:

* Objective cognitive impairments before hospital admission for the COVID-19 infection
* An unexpected incident leading to severe neurological damage after hospital discharge (such as stroke or traumatic brain injury)
* Contra-indications for MRI scanning (e.g. metal implants, cardiac pacemaker, claustrophobia, pregnancy, and tattoos in the head/neck region)
* Unwillingness to be informed about clinical relevant (abnormal) MRI-findings
* Contra-indications for a gadolinium-based MRI contrast agent (known allergy or insufficient kidney function determined by an eGFR < 30 mL/min)
* Physical inability to travel to one of the locations (e.g. bedridden patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of adult patients who survived a COVID-19 infection for which ICU hospital admission was necessary during the second/third pandemic wave (October 2020 - ongoing).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Radiological outcome | 12-24 months post ICU admission
  MRI abnormalities, focusing on vascular abnormalities and olfactory tractus (3T MRI), and lymphatics and the brainstem (7T MRI).
Neurological outcome | 12-24 months post ICU admission
  Residual neurological symptoms (including sense of smell/taste) and functional status.
Clinical outcome | 12-24 months post ICU admission
  severity of disease scores, (serial) factors of hyper coagulability and inflammation during ICU admission, neurological and cardiovascular (arterial/venous) complications during hospital admission.

SECONDARY OUTCOMES:
Neuropsychological outcome | 12-24 months post ICU admission
  Global deficits in cognitive and neurological functioning, objective changes in or loss of smell/taste, and residual signs of inflammation and hypercoagulability.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel JH Ariës, PhD/MD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided